CLINICAL TRIAL: NCT06109909
Title: A Novel Neurofeedback Intervention for Photosensitivity in Mild Traumatic Brain Injury
Brief Title: Pilot Study of Neurofeedback for Photosensitivity in Mild Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C4374-P
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Mild Traumatic Brain Injury; Photophobia
Keywords: photophobia; mild traumatic brain injury
MeSH Terms: conditions — Brain Concussion; Photophobia

STUDY DESIGN:
Intervention Model Description: After consent, participants will be randomly assigned to either the LIP-tES intervention or sham control group. Participants will complete 12 sessions over 6 weeks during which photosensitivity symptoms will be tracked using the Utah Photophobia Symptom Impact Scale (UPSIS). A subset of participants will also complete a resting-state MRI scan session during the initial visit and again during the 12th visit. A follow-up phone call will be placed after a 6 week wash-out period. Group assignment will be disclosed at this time and participants in the sham condition who would like to receive the LIP-tES intervention will be able to return for an additional 12 sessions over 6 weeks during which they will receive LIP-tES and photosensitivity symptoms will be tracked using the UPSIS questionnaire.
Who Masked: Participant
Masking Description: Sham treatment, single-blind design. During the sham treatment, we will prep and place electrodes in the same manner as participants receiving the LIP-tES treatment. However, no LIP-tES pulses will be sent from the system during the sham treatment. The operator will know which group the participant is assigned to but all aspects of study design and data collection will be the same from the perspective of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neurofeedback (Experimental): Half of the participants will be blindly assigned to receive 12 sessions of LIP-tES intervention over 6 weeks. A subset of these participants will also complete a resting-state MRI scan during the initial session (prior to LIP-tES intervention) and after their final LIP-tES intervention.
  Interventions: Device: Micro Current Neurofeedback Device using Low-Frequency Pulse-Based Transcranial Electrical Stimulation
- Sham Treatment (Sham Comparator): Half of the participants will be blindly assigned to receive 12 sessions of a sham intervention that will mirror all aspects of the LIP-tES intervention except that no neurofeedback pulses will be delivered. A subset of these participants will also complete a resting-state MRI scan at the beginning of the initial session and at the end of the 12th session.
  Interventions: Device: Micro Current Neurofeedback Device using Low-Frequency Pulse-Based Transcranial Electrical Stimulation

INTERVENTIONS:
Device: Micro Current Neurofeedback Device using Low-Frequency Pulse-Based Transcranial Electrical Stimulation — The EEG interface device is a J&J Engineering 1-330 C2 box. The software used to determine LIP-tES feedback patterns was developed by Neurogen High Performance Neurofeedback. The EEG sampling frequency is 256 Hz on each of 2 EEG acquisition channels. The feedback LIP-tES is delivered via the 4 EEG leads (A+,A-,B+,B-), with respect to the Common Neck Reference. During each session, 2 electrodes (A- and B-) are attached to the participant's left and right mastoids, while the remaining two electrodes (A+ and B+) are moved to various locations on the scale to record EEG signals. All four (A+,A-,B+,B-) electrodes are involved in applying weak electrical pulses back to the brain (feedback process). The brief feedback pulse (~100mV) is adaptive and determined based on the offset of the frequency spectrum recorded across the left and right hemisphere (A vs. B) electrodes in the time window immediately prior to stimulation.
  Other Names: LIP-tES intervention

SUMMARY:
The goal of this study is to complete a pilot study testing the feasibility and acceptability of low-intensity pulse-based transcranial stimulation (LIP-tES) neurofeedback intervention for reducing photosensitivity symptoms in Veterans with a history of mild traumatic brain injury (mTBI). The study will also complete resting-state MRI scans to assess neurophysiological markers of photosensitivity and changes associated with LIP-tES intervention.

DETAILED DESCRIPTION:
Photosensitivity (PS) is one of the more common sequelae of TBI, with over 50% of TBI patients reporting some level of PS in the acute and/or chronic stages. PS can range from mild to severe and can significantly impair social, physical, and cognitive functioning, as well as rehabilitation outcomes. While spectacle chromatic filters are conventionally used to alleviate symptoms, they are not designed to resolve issues with PS and have been associated with lower symptom recovery over time, underscoring the need to develop more effective, non-invasive treatment options that can reduce or eliminate PS. Recent work has shown that neurofeedback interventions, such as Low Intensity Pulse-Based Transcranial Electrical Stimulation (LIP-tES) may be effective in treating post-concussive symptoms and a preliminary case study from the investigators' research group suggests that LIP-tES may also be able to reduce PS symptoms in Veterans with a history of mild TBI. However, both the mechanism by which LIP-tES alters brain activity and alleviates symptoms across a range of disorders remains unclear as does the neurobiological basis of PS associated with mTBI and psychiatric comorbidities commonly seen in today's Veteran population. These knowledge gaps represent important limitations both for the clinical characterization of PS in Veterans and development/optimization of novel treatment options. This proposal will take an important first step in addressing these two important knowledge gaps. Aim 1: Complete a preliminary study testing the feasibility and acceptability of a novel LIP-tES intervention designed to reduce severity of PS in patients with a history of mTBI. Extending a recent case study completed by the investigators' research group, the investigators will complete a pilot study of LIP-tES for the treatment of PS in Veterans with a history of mTBI. The investigators will track recruitment capability (participants screened vs. enrolled, attrition rates and reasons for attrition), acceptability and suitability of the intervention, evaluate suitability of the sham procedure the investigators developed, and gain preliminary evaluation of participant responses to the intervention. Aim 2: Assess neurophysiological markers of PS and changes associated with LIP-tES intervention using resting-state fMRI. A subset of the participants will complete two MRI scans during the initial visit after the last LIP-tES or sham session. Preliminary work from the investigators' laboratory has identified a sparse connectome of regions that are predictive of moderate/severe PS ratings in a polymorbid sample of Veterans from the Translational Research Center for TBI and Stress Disorders (TRACTS) longitudinal cohort study. Extending this work, the investigators will test whether classification models using this previously identified connectome will correctly identify individuals who report a reduction in PS after treatment and whether connections are predictive of PS severity. By examining resting-state functional connectivity prior to and after completion of LIP-tES, the proposed study aims to increase the understanding of the underlying pathophysiological mechanisms of PS in mTBI and the mechanism by which LIP-tES may alleviate these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Documented history of mTBI at least 6 months prior to initial study visit
* Documented symptoms of photosensitivity
* Eye exam within the last 12 months documenting best-corrected acuity of 20/20 or better, normal pupillary function, color vision, no abnormalities on OCT scan, and normal Humphrey Visual Field test

Exclusion Criteria:

* History of strabismus or amblyopia
* Significant ocular media opacity that could reduce the amount of light entering the pupil in one or both eyes
* Previous or current history of retinal or optic nerve pathology in one or both eyes
* History of stroke and/or visual neglect
* History of neurodegenerative disease (e.g., Parkinson's, multiple sclerosis)
* History of epilepsy or seizures
* History of motor tics
* Current use of medications or substances that may severely affect pupillary response and/or increase photosensitivity
* Individuals with impaired decision-making capacity
* Illiterate or no English language proficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Utah Photophobia Symptom Impact Scale (UPSIS) | Baseline and again every two weeks through end of treatment, average of 6 weeks
  The UPSIS questionnaire is a 17-item questionnaire designed to quantitatively assess photosensitivity symptoms and their impact on activities of daily living. Scores range from 0-80 with higher values indicating more severe photosensitivity symptoms.

SECONDARY OUTCOMES:
Stimulation Related Sensations Questionnaire (SRSQ) | Baseline treatment visit
  The SRSQ will be administered to participants after the LIP-tES or sham session is complete. Results will be used to assess if participants report different sensations across conditions to examine if sham condition is appropriate control condition.
Change from Baseline in Neurobehavioral Symptom Inventory (NSI) | Baseline and again at study completion, an average of 6 weeks
  The NSI will be administered as a measure of general post-concussive symptoms
Change from Baseline in Headache Impact Test (HIT-6) | Baseline and again at study completion, an average of 6 weeks
  The HIT-6 will be administered to measure changes in headache frequency and severity over prior month.
Qualitative Assessment of Study Recruitment Capability | End of study data collection, approximately 2 years
  Qualitative assessment of ability to recruit participants into the study by examining recruitment rates and reported obstacles to recruitment over study period. Assessment will result in decision that recruitment capabilities are suitable or unsuitable for additional study with no change to targeted population with same inclusion/exclusion criteria.
Qualitative Assessment of Acceptability of Data Collection Methods | End of study data collection, approximately 2 years
  Qualitative assessment of the suitability of data collection procedures by examining the retention and follow-up rates as the participants moved through the study and intervention, adherence rates to study procedures, barriers to study participation reported by participants over the course of the study. Assessment will result in decision that current study protocol is suitable or unsuitable for additional study with no change to study design.
Change from Baseline in PTSD Checklist for DSM-5 (PCL-5) | Baseline and again at study completion, an average of 6 weeks
  The PCL-5 will be administered to measure changes in PTSD symptom severity.
Change from Baseline in Depression, Anxiety, and Stress Scale (DASS) | Baseline and again at study completion, an average of 6 weeks
  The DASS questionnaire will be administered to measure changes in severity of depression, anxiety, and stress symptoms.
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) | Baseline and again at study completion, an average of 6 weeks
  The PSQI will be administered to provide a measure of changes in global sleep quality.
Change from Baseline in Short Form McGill Pain Questionnaire | Baseline and again at study completion, an average of 6 weeks
  This questionnaire will be administered to provide a general measure of changes in chronic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca C Fortenbaugh, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No